CLINICAL TRIAL: NCT05645497
Title: Evaluation of the Efficacy and Safety of the FACET FIXation Implant Compared With Pedicle Screw Fixation in Patients With Degenerative Lumbar Spinal Stenosis.
Brief Title: Evaluation of the Efficacy and Safety of the FACET FIXation Implant.
Acronym: FACETFIX
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: SC Medica (Industry)
Responsible Party: Sponsor
Other Study IDs: 2022-A01783-40
Record Dates: First submitted 2022-12-01; First posted 2022-12-09 (Actual); Last update posted 2023-04-12 (Actual); Status verified 2023-04

CONDITIONS: Degenerative Lumbar Spinal Stenosis
MeSH Terms: interventions — Surgical Procedures, Operative; Pedicle Screws

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Patient with medical device FACET FIXATION: The FACET FIXATION group include all the patients with Lumbar Spinal Stenosis who underwent an open technique for decompression, specifically laminectomies, concomitant to FACET FIXATION from November 2017 (and having more than 2 years postop to date).
  Interventions: Procedure: Surgery with FACET FIXATION implants
- Patient with medical device Pedicle Screw: The Pedicle Screw group consiste of all the patients with Lumbar Spinal Stenosis who underwent an open technique for decompression, specifically laminectomies, concomitant to Pedicle Screw fixation from 2015 to 2016.
  Interventions: Procedure: Surgery with Pedicle Screw

INTERVENTIONS:
Procedure: Surgery with FACET FIXATION implants — Surgical treatment of degenerative lumbar spinal stenosis by lumbar decompression with FACET FIXATION implants
  Groups: Patient with medical device FACET FIXATION
Procedure: Surgery with Pedicle Screw — Surgical treatment of degenerative lumbar spinal stenosis by lumbar decompression with Pedicle Screw
  Groups: Patient with medical device Pedicle Screw

SUMMARY:
This is a single center, hybrid retrospective and prospective (ambispective) study to evaluate the safety and efficacy of the Facet Fixation implant.

The main objective is to evaluate the efficacy of the Facet Fixation implant compared with pedicle screw fixation to determine successful fusion in radiographic assessment at more than two years. Fusion is mainly defined as any sign of bony fusion between the facet joints or transverse processes when viewing the postoperative CT-scan at over 2 years.

DETAILED DESCRIPTION:
The primary endpoint is the successful fusion rate in radiographic assessment at more than 2 years.

ELIGIBILITY:
Inclusion Criteria:

* Patient is ≥ 18 years old at the time of the surgery
* The first back operation in the patient's life was for degenerative lumbar spinal stenosis
* Surgical treatment of degenerative lumbar spinal stenosis by lumbar decompression with Pedicle Screw fixation or FACET FIXation implant.
* Patient is able to understand the information related to the study
* Patient consents to participate to the clinical investigation and agrees (non-objection) on the use of his/her personal data.

Exclusion Criteria:

* Patient received FACET FIXation implant or Pedicle Screw fixation with supplemental interbody cages.
* Unilateral Pedicle Screw or FACET FIXation implant.
* Preoperative grade ≥II spondylolisthesis
* Preoperative scoliotic deviations >25°.
* Protected patient (under legal protection, deprived of liberty by judicial or administrative decision).
* Patient not covered by a social security scheme.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population will consist of adult patients diagnosed with degenerative lumbar spinal stenosis who underwent their first spinal operation for lumbar decompression with pedicle screws fixation or FACET FIXation implant from 2015 to 2020 (2015-2016 with Pedicle Screw and starting November 2017 with more than 2 years postop at the date of the visit with FACET FIXation implant).
Sampling Method: Probability Sample
Enrollment: 116 (Estimated)
Dates: Start 2023-01-17 (Actual); Primary Completion 2023-04-30 (Estimated); Study Completion 2023-04-30 (Estimated)

PRIMARY OUTCOMES:
The rate of fusion | 2 years
  The proportion of patients achieving the primary endpoint will be evaluated. The rate of fusion in the radiographic assessment is considered successful if all of the following criteria are achieved :
  * Evidence of bridging bone between the facet joints (Facet Fixation implant) or the transverse processes (pedicle screws) via computed tomography scan.
  * and ≤ 3mm translational motion between vertebrae on flexion / extension via dynamic X-rays.
  * and no evidence of lucency surrounding the device (≤25%).
  The main analysis will compare the successful fusion rate at 2+ years post-operative between the group with the Facet Fixation and the group with pedicle screws, by a confidence interval approach.

CONTACTS AND LOCATIONS:
Locations (1):
- Hôpitaux Civils de Colmar, Colmar, France

IPD SHARING:
Plan to Share IPD: No